CLINICAL TRIAL: NCT03460171
Title: The French hMPV Study: Clinical Features, Outcome and Prognosis of Human Metapneumovirus (hMPV) Lower Respiratory Tract Infections in Adult Inpatients
Brief Title: Clinical Features, Outcome and Prognosis of Human Metapneumovirus (hMPV) Lower Respiratory Tract Infections in Adult Inpatients
Acronym: French-hMPV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HAO 17024
Record Dates: First submitted 2017-12-11; First posted 2018-03-09 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Lower Resp Tract Infection; Human Metapneumovirus Infection
Keywords: Human Metapneumovirus; Paramyxoviridae infections; Lower-respiratory tract infections; Pneumonia
MeSH Terms: conditions — Paramyxoviridae Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The human metapneumovirus (hMPV) was first described in 2001. It belongs to the paramyxovirus family and is genetically close to the Respiratory Syncytial Virus (RSV). hMPV has a seasonal epidemic pattern, between January to April. Clinical symptoms of hMPV infection include influenza-like illness (fever, asthenia and curvatures) associated with signs of respiratory tract infection. The incidence of hMPV infection is higher in children than in adults. In child pneumonia, hMPV is the third most frequent isolated pathogen (14 % of the subjects), after rhinovirus and RSV. In hospitalized adults, hMPV was detected in 6 to 8% of the subjects with lower respiratory tract and in 4 % of subjects with pneumonia.

Clinical, radiological and biological features, as well as evolution course of hMPV infections have been mainly described in children. Clinical presentation of in adult seems polymorph, ranging from acute bronchitis or exacerbation of COPD to pneumonia. The frequency of viral-bacterial coinfection is unknown. Intensive care unit (ICU) admission may involve almost 1 for 10 patients. Elderly and immunocompromised subjects are probably high-risk subjects.

Currently, treatment of hMPV infections is mainly symptomatic. However, several anti-RSV drugs that are currently in clinical development have demonstrated an activity against other paramyxoviridae in pre-clinical studies. Consequently, it seems necessary to better characterize hMPV infections in adult inpatients: presentation, course profile and risk factors for morbidity and mortality. These data would help clinicians to identify high risk patients, and consequently to choose those who could benefit from coming treatments.

The French hMPV Study is observational prospective multicenter clinical study. The study population includes all consecutive adult inpatients with a community-acquired acute lower respiratory tract infection and a mPCR positive for hMPV on any respiratory sample. The primary objective is to describe the prognosis. The secondary objectives are i) to characterize clinical, radiological and biological features, ii) to describe the hospital course and the rate of ICU transfer; in ICU patients, to describe organ failures and supports, and iii) to describe the viral and/or bacterial coinfections. The primary endpoint is the number of subjects with a poor outcome (defined by the requirement for invasive mechanical ventilation and/or the death during the hospital stay).

DETAILED DESCRIPTION:
The human metapneumovirus (hMPV) was first described in 2001. It belongs to the paramyxovirus family (paramyxoviridae subfamily). hMPV is genetically close to the Respiratory Syncytial Virus (RSV). hMPV has a seasonal epidemic pattern, between January to April. Incubation period varies between 4 and 6 days. Clinical symptoms of hMPV infection are close to that of RSV, with influenza-like illness (fever, asthenia and curvatures) associated with signs of upper and/or lower respiratory tracts infection. The incidence of hMPV infection is higher in children than in adults. In a large cohort of children with respiratory illness or fever, hMPV was detected in 7 % of outpatients and 6 % of hospitalized children. The annual rate of hospitalization associated with hMPV infection has been estimated about 1 per 1000 children less than 5 years of age. In child pneumonia, hMPV is the third most frequent isolated pathogen (14 % of the subjects), after rhinovirus and RSV. In hospitalized adults, hMPV was detect in 6 to 8% of the subjects with a lower respiratory tract and in 4 % of subjects with a pneumonia.

Clinical, radiological and biological features, as well as evolution course of hMPV-associated infections have been mainly described in children. Clinical presentation of hMPV-associated infection in adult seems polymorph, ranging from acute bronchitis or exacerbation of chronic pulmonary diseases (COPD and asthma) to pneumonia. Viral-viral coinfections are not exceptional whereas the frequency of viral-bacterial coinfection is unknown. Intensive care unit (ICU) admission involved almost 1 for 10 patients. Elderly and immunocompromised subjects are probably high-risk subjects. Only one cohort of hMPV-infected patients admitted to ICU has been reported. Among the 40 patients, 6 were non-immunocompromised and without comorbidity. Factors associated with a poor prognosis were not studied.

Currently, treatment of hMPV-associated lower respiratory tract infections is mainly symptomatic. However, several anti-RSV drugs that are currently in clinical development in humans, have demonstrated an activity against other paramyxoviridae (hMPV and parainfluenza virus) in pre-clinical studies. These anti-RSV drugs should be available for clinicians in the next few years. Considering their activity against other paramyxoviridae, clinicians will probably attempt to use these anti-RSV drugs in non-RSV paramyxoviridae-associated lower respiratory tracts infections in adult inpatients. Consequently, it seems necessary to better characterize hMPV-associated lower respiratory tracts infections in adult inpatients: clinical, radiological and biological presentation, course profile and risk factors for morbidity and mortality. These data would help clinicians to identify high risk patients, and consequently to choose those who could benefit from coming treatments.

The French hMPV Study is observational prospective multicenter clinical study. The study population includes all consecutive adult inpatients with a community-acquired acute lower respiratory tract infection and a mPCR positive for hMPV on any respiratory sample. The primary objective is to describe the prognosis. The secondary objectives are i) to characterize the clinical (time from onset to hospital admission, general symptoms, respiratory symptoms and signs), radiological and biological features, ii) to describe the hospital course and the rate of ICU transfer; in ICU patients, to describe organ failures and supports, and iii) to describe the viral and/or bacterial coinfections.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) inpatients with:
* an acute lower respiratory tract infection, defined by the presence of two of the following criteria in the 5 days preceding hospital admission or during the present hospital stay : fever, cough, expectoration, exercise or rest dyspnea, crackles, tubal breath, signs of respiratory failure (respiratory rate higher than 30 per minute...), thoracic pain, oxygen therapy, mechanical ventilation;
* a respiratory mPCR (upper respiratory tracts specimen such as nasopharyngeal swab or lower respiratory tract specimen such as tracheal or bronchial aspiration or bronchoalveolar lavage) positive for hMPV in the 5 days following hospital admission.

Exclusion Criteria:

* Patient already included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients admitted to hospital with an acute lower respiratory tract infection and a respiratory MPCR positive for hMPV.
  Participating centres are respiratory diseases departments, infectious diseases departments and intensive care units of secondary and tertiary care hospitals in France.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the number of subjects with a poor outcome (defined by the requirement for invasive mechanical ventilation and/or the death during the hospital stay or at 60 days). | during the hospital stay or at 60 days

SECONDARY OUTCOMES:
Age (years) | at hospital admission
Gender (H or F) | During the first 24 hours of ICU stay
Height (cm) | During the first 24 hours of ICU stay
Weight (kg) | During the first 24 hours of ICU stay
Charlson score (points) | During the first 24 hours of ICU stay
Presence or absence of each of the following comorbidities | During the first 24 hours of ICU stay
  smoking, asthma, COPD, chronic respiratory insufficiency requiring long term oxygen therapy, diabetes, hypertension, chronic heart failure NYHA III IV, coronary artery disease, cerebral arterial disease, chronic dialysis and cirrhosis Child Pugh B-C
Presence or absence of each of the following immunocompromised conditions | During the first 24 hours of ICU stay
  HIV infection, splenectomy, long term steroid therapy, other long term immunosuppressive drug, anticancer agents, solid organ transplant, cancer or hematologic neoplasm
Presence or absence of each of the following factors of health-care associated lower respiratory tract infection | During the first 24 hours of ICU stay
  hospitalization for ≥ 2 days in the preceding 90 days and institutionalization
Antipneumococcal and anti-flu vaccine | During the first 24 hours of ICU stay
Date of first respiratory symptoms (date) | During the first 24 hours of ICU stay
Respiratory rate (maximum) during the first 24 hours of hospital stay (/min) | During the first 24 hours of ICU stay
Temperature (maximum) during the first 24 hours of hospital stay (°C) | During the first 24 hours of ICU stay
Heart rate (maximum) during the first 24 hours of hospital stay (/min) | During the first 24 hours of ICU stay
Glasgow score (minimum) during the first 24 hours of hospital stay (points) | During the first 24 hours of ICU stay
Blood leucocytes (maximum) at hospital admission (G/L) | During the first 24 hours of ICU stay
Blood neutrophils (maximum) at hospital admission (G/L) | During the first 24 hours of ICU stay
Blood lymphocytes (maximum) at hospital admission (G/L) | During the first 24 hours of ICU stay
Blood platelets (maximum) at hospital admission (G/L) | During the first 24 hours of ICU stay
Partial pressure of O2 (mmHg) | During the first 24 hours of ICU stay
Number of quadrant with radiological abnormalities on the Chest X-Ray (number, maximum=4) | During the first 48 hours of ICU stay
Viral co-infection | During Hospital stay, censored at 60 days
Bacterial co-infection | During Hospital stay, censored at 60 days
Duration of mechanical ventilation support (invasive or non invasive) | during hospital stay or at 60 days
Shock (vasopressor support) | during hospital stay or at 60 days
ARDS (Berlin definition) | during hospital stay or at 60 days
Duration of ICU stay | during hospital stay or at 60 days
Duration of hospital stay (days) | censored at 60 days
Death | during hospital stay or at 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Voiriot, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Muriel Fartoukh, MD PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de réanimation-Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: No